CLINICAL TRIAL: NCT00836030
Title: DiabCare Asia 2008. A Cross-Sectional Survey to Evaluate Diabetes Management, Control, Complications, Psychosocial Aspects of Diabetic Patients in Asia and To Evaluate Perceptions and Practices of Physicians and Patients About Diabetes Management in Asia
Brief Title: A Survey to Evaluate Diabetes Management, Control, Chronic Complications, Psychosocial Aspects of Diabetic Subjects in Singapore
Acronym: DiabCare Asia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3710
Record Dates: First submitted 2009-01-30; First posted 2009-02-04 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate current status of diabetes management, control and complications in diabetic subjects in Asia.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients registered in the particular centre for more than 12 months
* Patients should have visited the centre at least once in the last 3-6 months apart from the initial visit
* Patients willing to sign informed consent form

Exclusion Criteria:

* Repetition of any patient as patients should not be included twice for any reason
* Unwilling to participate or unable to comply with protocol requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus (both type 1 and type 2) being treated at general hospitals, diabetes clinics and referral clinics will be selected according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 854 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Mean age of onset of type 1 and 2 diabetes mellitus | at baseline visit/study start
Mean duration of treatment of type 2 DM | at baseline visit/study start
Percentage of patients on Insulin and OAD therapy | at baseline visit/study start
Mean duration of diabetes in type 1 and type 2 patients respectively | at baseline visit/study start
Mean FPG and PPG of diabetic patients | at baseline visit/study start
Mean HbA1c of diabetic patients | at baseline visit/study start
Percentage of diabetic patients with HbA1c target below or equal to 7.0% | at baseline visit/study start
Percentage of diabetic patients with HbA1c target below or equal to 6.5% | at baseline visit/study start
Percentage of diabetic patients having dyslipidemia and hypertension | at baseline visit/study start
Percentage of diabetic patients having cardiovascular complications | at baseline visit/study start
Percentage of diabetic patients having peripheral vascular disease | at baseline visit/study start
Percentage of diabetic patients having diabetic nephropathy | at baseline visit/study start
Percentage of diabetic patients having diabetic eye complications | at baseline visit/study start

SECONDARY OUTCOMES:
Patients' perception will be analysed through Patient questionnaire measuring - Psychological well-being, Quality of life, Patients' compliant to treatment | at baseline visit/study start
Physician perception of diabetes and its management will be analysed through Physician questionnaire measuring awareness about - HbA1c test and its goal, Anti-diabetic treatment, Barriers towards optimum diabetes control | at baseline visit/study start
Duration of diabetes associated with highest number of diabetic complications | at baseline visit/study start
Minimum duration of diabetes associated with 10% incidence of diabetic complications (CVD, Nephropathy and retinopathy) | at baseline visit/study start

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Singapore, Singapore

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com